CLINICAL TRIAL: NCT07062562
Title: The Effect of Repeated Sessions of Whole-body Neuromuscular Electrical Stimulation (NMES), With or Without Subsequent Intake of a Protein Bolus, on Muscle Protein Synthesis in Healthy, Young Volunteers During 3 Days of Bed Rest
Brief Title: The Effect of Repeated Whole-body NMES Sessions With or Without Protein Intake on Muscle Protein Synthesis During 3 Days of Bed Rest in Healthy Young Volunteers
Acronym: SPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Marlou Dirks, Assistant Professor, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL88628.028.24
Record Dates: First submitted 2025-05-22; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Muscle Wasting
Keywords: NMES; Skeletal Muscle Metabolism; Protein; Disuse
MeSH Terms: conditions — Muscular Atrophy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled intervention trial with three parallel groups. Participants will undergo 3 days of bed rest and receive either sham-NMES, whole-body NMES, or whole-body NMES with protein to assess the effects on muscle protein synthesis. The study will measure muscle protein metabolism, strength, and function to determine whether NMES and protein intake can mitigate muscle loss during immobilization.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Sham Comparator): Sham-NMES with standard nutrition
  Interventions: Other: Sham (No Treatment); Other: Standard nutrition
- Whole-body NMES group (Active Comparator): Whole-body NMES stimulation with standard nutrition
  Interventions: Other: NMES; Other: Standard nutrition
- Whole-body NMES + protein group (Active Comparator): Whole-body NMES with a 20g protein bolus on top of the standard nutrition
  Interventions: Other: NMES; Dietary Supplement: Protein bolus (20g); Other: Standard nutrition

INTERVENTIONS:
Other: Sham (No Treatment) — A placebo treatment in which no actual electrical stimulation is delivered, serving as a control for the active NMES.
  Arms: Control group
Other: NMES — Active neuromuscular electrical stimulation applied to the entire body to induce muscle contractions through small electric currents.
  Arms: Whole-body NMES + protein group; Whole-body NMES group
Dietary Supplement: Protein bolus (20g) — A bolus dose of 20 grams of protein provided after the NMES intervention to assess the combined effect of muscle stimulation and protein intake on muscle protein metabolism.
  Arms: Whole-body NMES + protein group
Other: Standard nutrition — Provision of a normal Western standardized diet.

SUMMARY:
The goal of this clinical trial is to examine the effect of whole-body electrostimulation with protein intake on muscle protein synthesis, muscle mass and function during bed rest in healthy young adults (18-35 years). The main questions to answer are:

* Does whole-body NMES followed by protein intake improve muscle protein synthesis rates during 3 days of bed rest?
* Does repeated NMES sessions offer protective effects on muscle mass and function during extended periods of inactivity?

Researchers will compare sham electrical electrostimulation, electrical stimulation and electrical stimulation + protein groups to see if whole-body electrostimulation combined with protein intake offers the greatest improvement in muscle protein metabolism and muscle preservation.

Participants will:

* Undergo 3 days of bed rest while receiving one of the following interventions:

  * Sham-NMES followed by standard nutrition (CON)
  * Whole-body NMES followed by standard nutrition(NMES)
  * Whole-body NMES followed by a bolus of 20g protein (NMES+PRO)
* Receive heavy water (D2O) to assess body water turnover.
* Undergo leg extension exercises to assess muscle function.
* Have quadriceps muscle thickness measured via ultrasound.
* Provide saliva samples for analysis.
* Have calf circumference measured to monitor changes in muscle mass.

DETAILED DESCRIPTION:
Patients admitted to the hospital often experience prolonged bed rest, which can lead to rapid muscle loss and weakness. In the intensive care unit (ICU), this condition, known as ICU-acquired weakness (ICU-AW), affects up to 50% of patients and can lead to longer mechanical ventilation times, increased morbidity, and a reduced quality of life after hospital discharge. One of the key reasons for muscle loss during bed rest is an impaired response to dietary protein, which normally helps maintain muscle mass.

Neuromuscular electrical stimulation (NMES) is a method that uses small electrical currents to stimulate muscle contractions, potentially counteracting muscle loss during periods of inactivity. Previous research has shown that NMES applied to the quadriceps muscles can reduce muscle loss in sedated patients and improve muscle protein synthesis in individuals with type 2 diabetes. However, the effects of whole-body NMES in combination with timed protein intake on muscle protein metabolism during bed rest are still unknown.

This study aims to investigate the impact of both a single session and repeated sessions of whole-body NMES, with or without subsequent protein intake, on muscle protein synthesis rates, muscle mass, and function during 3 days of bed rest in healthy young adults.

Study Design:

This is a randomized, placebo-controlled clinical trial with three parallel groups. Participants will be randomly assigned to one of the following groups:

* Control Group (CON): Sham-NMES + standard nutrition
* NMES Group (NMES): Whole-body NMES + standard nutrition
* NMES + Protein Group (NMES+PRO): Whole-body NMES + 20g protein bolus

Study Procedures:

Participants will be healthy adults (18-35 years, male and female) and will undergo the following procedures:

* 3 days of strict bed rest to simulate hospitalization-related muscle disuse
* Neuromuscular electrical stimulation (NMES) sessions to assess its effect on muscle metabolism
* Muscle biopsies to measure changes in muscle protein synthesis at the molecular level
* Consumption of deuterium oxide (D₂O or "heavy water") to track muscle protein turnover
* Multiple blood and saliva samples to analyze protein metabolism markers
* Leg extension tests to assess changes in muscle function
* Quadriceps muscle thickness measurements via ultrasound
* Calf circumference measurements to assess muscle mass changes

This study will provide critical insights into how NMES and protein intake can help counteract muscle loss and weakness during hospitalization and may contribute to the development of more effective rehabilitation strategies for ICU and bedridden patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18-35 years
* 18.5 < BMI < 30 kg·m2
* Recreationally active (performing non-competitive physical exercise at least one time per week for minimally 30 minutes)

Exclusion Criteria:

* Employed or undertaking a thesis or internship at the department of Human and Animal Physiology at Wageningen University
* Smoking
* Diabetes (Type 1, Type 2, or genetic form of diabetes)
* Any diagnosed cardiovascular (heart) disease or high blood pressure (≥140 mmHg systolic and/or

  ≥90 mmHg diastolic)
* Chronic use of any prescribed or over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices)
* Known allergy to lidocaine
* Prone to keloid forming (i.e. hyperplastic growth of scars)
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g.

arthritis, spasticity/rigidity, all neurological disorders and paralysis)

* Regular use of dietary protein and/or amino acid supplements (>3 times per week)
* Currently involved in a structured progressive resistance training programme (>3 times per week)
* A personal or family history of thrombosis (clots), epilepsy, seizures, or schizophrenia
* Any previous motor disorders or disorders in muscle and/or lipid metabolism
* Any back, leg, knee, neck, shoulder or postural complaints
* Presence of an ulcer in the stomach or gut and/or strong history of indigestion
* Contra-indications for DXA scans (e.g. undergoing radiologic examination)
* Lactose intolerance
* Known severe kidney problems
* Pregnant or breastfeeding
* Unable to give consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative myofibrillar fractional synthesis rate | Habitual MPS (Day -2 to Day 0), Acute effect of NMES (+protein bolus) (0 hours to 5 hours on Day 0), Bedrest MPS (Day 0 to Day 3),
  A measure of muscle protein synthesis between two given time points.

SECONDARY OUTCOMES:
Quadriceps Muscle Layer Thickness | Between Day -21 and Day -5, Day 0, Day 3, Day 6, Week 6
  Assessed using ultrasound, this measures changes in muscle size, indicating muscle loss or preservation during bed rest and NMES intervention.
Body Composition | Day 0 and Day 3.
  Evaluates muscle mass to determine overall changes.
Body composition | Time Frame: Day 0 and Day 3.
  Evaluates fat distribution to determine overall changes.
Quadriceps Muscle Function | Between Day -21 and Day -5, Day 0, Day 3, Day 6, Week 6
  Assessed via a leg dynamometer.
Quadriceps Muscle Strength | Between Day -21 and Day -5, Day 0, Day 3, Day 6, Week 6
  Assessed via a leg dynamometer.
Handgrip Strength | Between Day -21 and Day -5, Day 0, Day 3, Day 6, Week 6
  Assessed via a hand dynamometer.
Whole-Body Nitrogen Balance | Day 0 to Day 3
  The balance between nitrogen intake (from dietary protein) and nitrogen loss (through urine and other excretions)

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands